CLINICAL TRIAL: NCT01418352
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Safety and Efficacy of Fixed-Dose Once-weekly Oral Aripiprazole in Children and Adolescents With Tourette's Disorder
Brief Title: Efficacy & Safety Study of Once-weekly Oral Aripiprazole in Children and Adolescents With Tourette's Disorder (TD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 31-10-273
Record Dates: First submitted 2011-08-01; First posted 2011-08-17 (Estimated); Results first posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Tourette's Disorder
Keywords: Tourette's Disorder; Tic disorders
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Matching Placebo (Placebo Comparator): Participants received aripiprazole matching placebo, tablets, orally, once weekly for 8 weeks in the Double-blind Treatment Period.
  Interventions: Drug: Placebo
- Aripiprazole 52.5 mg (Experimental): Participants received aripiprazole 52.5 mg, tablets, orally, once weekly for 8 weeks in the Double-blind Treatment Period.
  Interventions: Drug: Aripiprazole
- Aripiprazole 77.5 mg (Experimental): Participants received aripiprazole 77.5 mg, tablets, orally, once weekly for 8 weeks in the Double-blind Treatment Period.
  Interventions: Drug: Aripiprazole
- Aripiprazole 110 mg (Experimental): Participants received aripiprazole 110 mg, tablets, orally, once weekly for 8 weeks in the Double-blind Treatment Period.
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Aripiprazole tablets once weekly for 8 weeks.
  Other Names: ABILIFY
  Arms: Aripiprazole 110 mg; Aripiprazole 52.5 mg; Aripiprazole 77.5 mg
Drug: Placebo — Aripiprazole matching-placebo once-weekly for 8 weeks.
  Arms: Matching Placebo

SUMMARY:
The goal of the current trial is to determine efficacy and safety of once-weekly aripiprazole in reducing Total Tic Severity (TTS) score in children and adolescents with Tourette's Disorder.

ELIGIBILITY:
Inclusion Criteria:

* 7 to 17 year old with diagnostic and statistical manual of mental disorders, fourth edition -text revision (DSM-IV-TR) diagnostic criteria for Tourette's disorder (TD), confirmed by the kiddie schedule for affective disorders and schizophrenia - present and lifetime version (K-SADS-PL), including the Diagnostic Supplement 5
* Has a total tic score (TTS) ≥20 on the yale global tic severity scale (YGTSS) at Screening and Baseline
* Presenting tic symptoms cause impairment in the participant's normal routines, which include academic achievement, occupational functioning, social activities, and/or relationships
* Females of childbearing potential must have a negative pregnancy test, must be practicing acceptable double-barrier methods of contraception, and must not be pregnant or lactating.
* Written informed consent form (ICF) obtained from a legally acceptable representative & informed assent at Screening as applicable by study center's Institutional review board/independent ethics committee (IRB/IEC)
* The participant, designated guardian(s) or caregiver(s) are able to comprehend and satisfactorily comply with the protocol requirements, as evaluated by the investigator.

Exclusion Criteria:

* Clinical presentation and/or history, consistent with another neurologic condition that may have accompanying abnormal movements.
* History of schizophrenia, bipolar disorder, or other psychotic disorder.
* Participant receiving psychostimulants for treatment of attention-deficit disorder/Attention-deficit hyperactivity disorder (ADD/ADHD) and who have developed and/or had exacerbations of tic disorder after initiation of stimulant treatment.
* Currently meets DSM-IV-TR criteria for a primary mood disorder.
* Severe obsessive-compulsive disorder (OCD), per children's yale-brown obsessive compulsive scale (CY-BOCS) score >16.
* Taken aripiprazole within 30 days of the Screening visit.
* Received any investigational agent in a clinical trial within 30 days prior to Screening or who were randomized into a clinical trial with Once-weekly aripiprazole at any time.
* History of neuroleptic malignant syndrome.
* Sexually active participants not using 2 approved methods of contraception; breastfeeding or pregnant.
* Risk of committing suicide
* Bodyweight lower than 16 kg
* Taken neuroleptic or antiparkinson drugs <14 days prior to randomization.
* Requiring cognitive-behavioral therapy (CBT) for TD during study.
* Participant meets DSM-IV-TR criteria for any significant psychoactive substance use disorder within the past 3 months.
* Positive drug screen
* Participant requires medications not allowed per protocol
* Use of CYP2D6 and CYP3A4 inhibitors or CYP3A4 inducers within 14 days prior to dosing and for duration of study.
* Inability to swallow tablets or tolerate oral medication
* Abnormal laboratory test results, vital signs and Electrocardiogram (ECG) results

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2011-08-02 (Actual); Primary Completion 2014-03-12 (Actual); Study Completion 2014-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Kohegyi, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (31):
- United States (12):
  - Dothan, Alabama
  - San Francisco, California
  - Gainesville, Florida
  - Miami, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Omaha, Nebraska
  - Manhasset, New York
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Charlottesville, Virginia
  - La Crosse, Wisconsin
- Bulgaria (3):
  - Rousse
  - Sofia
  - Varna
- Germany (5):
  - Aachen
  - Dresden
  - Hanover
  - München
  - Ulm
- Romania (4):
  - Bucharest
  - Cluj-Napoca
  - Craiova
  - Iași
- Ukraine (7):
  - Donetsk
  - Kharkiv
  - Kyiv
  - Luhansk
  - Poltava
  - Stepanovka
  - Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/.
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 105 participants were screened and 83 were randomized to the treatment. The randomized participants were recruited at 38 sites in the following 5 countries: Bulgaria, Germany, Romania, Ukraine, and the US.
Pre-assignment Details: This study consisted of 2 distinct phases: a Pre-treatment Phase and a Treatment Phase. The Pre-treatment Phase consisted of a Screening period, a Washout period, and a Baseline visit. This was followed by an 8-week Treatment Phase. There was a follow-up period (30 days) for those participants who did not roll-over into the Open-label Study 31-10-274 (NCT01416441).
Groups:
- Aripiprazole 52.5 mg: Participants received aripiprazole 52.5 mg, tablet, orally, once weekly for the 8-week Double-blind Treatment Period.
- Aripiprazole 77.5 mg: Participants received aripiprazole 77.5 mg, tablet, orally, once weekly for the 8-week Double-blind Treatment Period.
- Aripiprazole 110 mg: Participants received aripiprazole 110 mg, tablet, orally, once weekly for the 8-week Double-blind Treatment Period.
- Matching Placebo: Participants received aripiprazole matching placebo, tablets, orally, once weekly for the 8-week Double-blind Treatment Period.
Period: Overall Study
Arm/Group | Aripiprazole 52.5 mg | Aripiprazole 77.5 mg | Aripiprazole 110 mg | Matching Placebo
Started | 20 | 21 | 21 | 21
Completed | 17 | 17 | 16 | 18
Not Completed | 3 | 4 | 5 | 3
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Sponsor Discontinued Trial Site | 0 | 2 | 2 | 2
Not completed — Subject Withdrew Consent | 0 | 1 | 2 | 1
Not completed — Protocol Deviation | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy as Determined by the Investigator | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Intention-to-Treat (ITT) Sample included participants randomly assigned to the double-blind treatment (regardless of whether or not they were dosed with study drug).
Groups:
- Matching Placebo: Participants received aripiprazole matching placebo tablets, orally, once weekly for the 8-week Double-blind Treatment Period.
- Total: Total of all reporting groups
Arm/Group | Aripiprazole 52.5 mg | Aripiprazole 77.5 mg | Aripiprazole 110 mg | Matching Placebo | Total
Number analyzed (Participants) | 20 | 21 | 21 | 21 | 83
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.5 (3.4) | 11.7 (2.8) | 12.5 (2.7) | 11.8 (2.7) | 11.9 (2.9)
Age, Customized [Count of Participants; unit: Participants]
  7 to 12 years | 12 | 11 | 11 | 14 | 48
  13 to 17 years | 8 | 10 | 10 | 7 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 3 | 6 | 20
  Male | 17 | 13 | 18 | 15 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 2 | 5
  Not Hispanic or Latino | 20 | 19 | 20 | 19 | 78
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 12 | 19 | 19 | 19 | 69
  Black or African American | 8 | 2 | 2 | 2 | 14
Weight [Mean (Standard Deviation); unit: Kilogram] | 44.7 (16.3) | 49.0 (16.2) | 52.8 (19.6) | 45.0 (12.5) | 47.9 (16.4)
Height [Mean (Standard Deviation); unit: centimeter] | 148.5 (19.0) | 151.8 (16.5) | 157.5 (14.8) | 151.8 (14.4) | 152.4 (16.3)
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kilogram per meter squared (kg/m^2)] | 19.6 (3.7) | 20.7 (3.8) | 20.6 (4.9) | 19.3 (3.7) | 20.0 (4.0)
Time since first diagnosis for Tourette's Disorder [Mean (Standard Deviation); unit: years] — Time since first diagnosis for Tourette's Disorder (years) = (date of screening assessment - date of first diagnosis + 1)/365.25
  years | 3.5 (3.0) | 1.8 (2.5) | 3.0 (3.5) | 2.6 (2.3) | 2.7 (2.9)
Yale Global Tic Severity Scale Total Tic Score (YGTSS TTS) [Mean (Standard Deviation); unit: score on a scale] — The YGTSS is a semi-structured clinical interview designed to measure the tic severity. This scale consisted of a tic inventory, with 5 separate rating scales to rate the severity of symptoms, and an impairment ranking. Ratings were made along 5 different dimensions on a scale of 0 to 5 for motor and vocal tics, each including number, frequency, intensity, complexity, and interference. The YGTSS TTS was the summation of the severity scores of motor and vocal tics. The total tic score (TTS) ranged from 0 (none) to 50 (severe).
  score on a scale | 28.2 (5.6) | 30.1 (5.8) | 31.4 (6.7) | 31.1 (5.5) | 30.2 (6)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Week 8 in Yale Global Tic Severity Scale (YGTSS) Total Tic Score
Description: The YGTSS is a semi-structured clinical interview designed to measure the tic severity. This scale consisted of a tic inventory, with 5 separate rating scales to rate the severity of symptoms, and an impairment ranking. Ratings were made along 5 different dimensions on a scale of 0 to 5 for motor and vocal tics, each including number, frequency, intensity, complexity, and interference. The YGTSS TTS was the summation of the severity scores of motor and vocal tics. The total tic score (TTS) ranged from 0 (none) to 50 (severe) with higher score represent more severe symptoms (greater reduction from baseline for greater improvement).
Time Frame: Baseline and Week 8
Population: The Intention-to-Treat (ITT) Sample included participants randomly assigned to the double-blind treatment (regardless of whether or not they were dosed with study drug). Overall number of participants analyzed are participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Aripiprazole 52.5 mg | Aripiprazole 77.5 mg | Aripiprazole 110 mg | Matching Placebo
Number analyzed (Participants) | 17 | 17 | 16 | 18
score on scale | -8.2 (4.8) | -9.9 (6.7) | -14.5 (7.7) | -9.6 (7.5)

2. Secondary Outcome: Mean Change From Baseline in Clinical Global Impressions Scale for Tourette's Syndrome (CGI-TS) Score
Description: The severity of illness and efficacy of study medication for each participant were rated using the CGI-TS scale. The study physician rated the participants total improvement whether or not it is due to study treatment. All responses were compared to the participants condition at Baseline (Day 0). Response choices include: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Aripiprazole 52.5 mg | Aripiprazole 77.5 mg | Aripiprazole 110 mg | Matching Placebo
Number analyzed (Participants) | 17 | 17 | 16 | 18
score on scale | -0.9 (0.6) | -1.1 (0.9) | -1.3 (1.0) | -1.0 (0.9)

3. Secondary Outcome: Mean Change From Baseline in Gilles de la Tourette Quality of Life (GTS-QOL) Overall Score at Week 8
Description: The GTS-QOL is a disease-specific patient-reported scale for the measurement of health-related quality of life in participants with Tourette's Disorder, taking into account the complexity of the clinical picture of the disease. The questionnaire consists of a 27-item Tourette's Disorder-specific scale with 4 subscales (psychological, physical, obsessional, and cognitive). The GTS-QOL total score ranged from 0 (extremely dissatisfied with life) and 100 (extremely satisfied with life). A positive change from Baseline indicates improvement.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Aripiprazole 52.5 mg | Aripiprazole 77.5 mg | Aripiprazole 110 mg | Matching Placebo
Number analyzed (Participants) | 17 | 17 | 16 | 18
score on scale | 8.8 (14.1) | 3.8 (24.4) | 13.1 (20.9) | 13.4 (15.9)

ADVERSE EVENTS:
Time Frame: From first dose up to 30 days post last dose (Up to approximately 12 weeks)
Groups:
- Aripiprazole 77.5 mg: Participants received aripiprazole 77.5 mg, tablet, orally once weekly for the 8-week Double-blind Treatment Period.
- Aripiprazole 110 mg: Participants received aripiprazole 110 mg, tablet, orally once weekly for the 8-week Double-blind Treatment Period.
Arm/Group | Aripiprazole 52.5 mg | Aripiprazole 77.5 mg | Aripiprazole 110 mg | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 8/20 | 4/21 | 16/21 | 4/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole 52.5 mg (N=20) | Aripiprazole 77.5 mg (N=21) | Aripiprazole 110 mg (N=21) | Matching Placebo (N=21)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Drug Prolactin Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight Increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 8 (8) | 2 (2)
Sedation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 3 (3) | 6 (6) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations of the trial such as small numbers of subjects analyzed or technical problems leading to unreliable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.